CLINICAL TRIAL: NCT04794569
Title: Tinzaparin Lead-In to Prevent the Post-Thrombotic Syndrome Phase IV Pilot Study
Brief Title: Tinzaparin Lead-In to Prevent the Post-Thrombotic Syndrome
Acronym: TILE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: funding discontinued
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: LEO Pharma (Industry); Sunnybrook Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3315
Record Dates: First submitted 2021-02-24; First posted 2021-03-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-06

CONDITIONS: Deep Vein Thrombosis; Post Thrombotic Syndrome
Keywords: tinzaparin
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Tinzaparin; Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients will be instructed not to disclose their treatment to PTS assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tinzaparin (Experimental): initial 3-week lead-in course of low molecular weight heparin (tinzaparin 175 units/Kg sc daily) followed by a direct oral anticoagulant (rivaroxaban 20mg po daily) for at least 3 months
  Interventions: Drug: tinzaparin
- Rivaroxaban (Active Comparator): Direct oral anticoagulant only (rivaroxaban 15mg po BID for 3 weeks followed by rivaroxaban 20mg po daily ) for at least 3 months
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: tinzaparin — low molecular weight heparin
  Arms: Tinzaparin
Drug: Rivaroxaban — direct oral anticoagulant
  Arms: Rivaroxaban

SUMMARY:
The TILE pilot study will be a multicenter, open-label, assessor-blinded RCT (randomized control trial) comparing extended LMWH (Low Molecular Weight Heparin) vs. DOAC (Direct Oral Anticoagulants) to PTS (prevent post thrombotic syndrome) in patients with DVT (Deep Vein Thrombosis).

DETAILED DESCRIPTION:
The TILE pilot study will investigate the magnitude of difference in effectiveness between LMWH (low molecular weight heparin, tinzaparin) plus DOAC (Direct Oral Anticoagulants, rivaroxaban) vs. DOAC alone to determine the sample size and assess feasibility for a larger study assessing the effectiveness of an initial 3-week lead-in course of LMWH (tinzaparin) compared to DOAC alone (rivaroxaban) in patients with proximal DVT (Deep Vein Thrombosis) at high risk of developing PTS (Post-Thrombotic Syndrome). PTS is a frequent, costly and burdensome complication of DVT, especially for patients with iliac or femoral vein DVT who have a high risk of developing PTS and severe PTS. Anticoagulant therapy appears to influence this risk, with a higher frequency of PTS in patients with DVT who receive suboptimal treatment with a VKA (Vitamin K Antagonist). DOAC are expected to avoid this and other limitations of VKA therapy and have become the standard of care for patients with DVT. Extended treatment of DVT with LMWH, by providing more effective anticoagulation and by reducing inflammation, appears to restore venous patency and reduce venous reflux compared to VKA and probably to DOAC. Extended treatment of DVT with LMWH, therefore, has the potential to reduce PTS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with objectively confirmed acute (i.e. onset of symptoms <10 days) symptomatic iliac or common femoral DVT (DVT diagnosis will be made with a Compression Ultrasound (CUS) according to standardized consensus criteria)

Exclusion Criteria:

1. Age < 18 years
2. History of ipsilateral DVT (distal and/or proximal)
3. Active cancer
4. Thrombolysis or other invasive early thrombus removal technique to treat DVT or PE
5. Pregnant or breast feeding
6. Impaired renal function (creatinine clearance < 30 ml/min according to Cockcroft-Gault formula)
7. Concomitant use of drugs that interact with rivaroxaban (i.e. keto- or itraconazole, ritonavir)
8. Allergy or hypersensitivity to heparin or rivaroxaban, including heparin induced thrombocytopenia
9. Anticoagulant therapy contraindicated because of presence of active bleeding or condition with high risk of bleeding (e.g. peptic ulcer, acute or subacute septic endocarditis, uncontrolled severe hypertension, other)
10. Thrombocytopenia (platelet count < 100 x 109/L)
11. Liver disease (including Child-Pugh Class B and Class C) associated with coagulopathy
12. Body weight > 120 kg or < 40 kg
13. Need for treatment with daily NSAIDs or antiplatelet agent (ibuprofen < 1200 mg/day, aspirin ≤ 160 mg/day or clopidogrel ≤ 75 mg/day are permitted)
14. Treatment with therapeutic doses of anticoagulants for > 72 hours
15. Mechanical heart valve
16. Antiphospholipid syndrome
17. Sulphite sensitivity
18. Lactose sensitivity
19. Life expectancy < 1 year
20. Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
PTS at 6 months | 6 months post randomization
  Proportion of patients with PTS at 6 months using the Villalta scale. PTS will be diagnosed using the Villalta scale. This clinical scale is the recommended standard to diagnose PTS.
Main feasibility | 3 months post randomization
  Main feasibility outcomes: a. Proportion of eligible patients, among patients screened b. Proportion of recruited patients, among patients who are eligible c. Proportion of patients who are compliant with tinzaparin, among recruited patients assigned to tinzaparin arm.

SECONDARY OUTCOMES:
PTS severity | 6 months post randomization
  The Villalta scale will be used to grade the severity of PTS (mild, moderate, severe) at 6 months post randomization.
Villalta score at 10 days | 10 days post randomization
  Villalta score at 10 days
DVT-related leg pain | Two time points: at 10 days and at 3 months post randomization
  DVT-related leg pain will be assessed using an 11-point Likert rating scale (0 no pain, 10, worst possible pain, during the last 24 hours). This relates to sub-acute DVT pain and not a pain that could have been caused by LMWH injection
Global Improvement | Two time points: at 10 days and at 3 months post randomization
  Assessing Patient's global improvement using the Patient's global improvement scale (On a scale of 1 to 7, where 1 is extremely improved and 7 is extremely deteriorated).
Patient's satisfaction with treatment | Two time points: at 3 weeks and at 6 months post randomization
  Patient's satisfaction with treatment and patient's global improvement will be assessed using a 7-point Likert visual analog scale questionnaire (1 = extremely satisfied to 7 = extremely dissatisfied).
QOL (Quality of Life) score - SF-36 | Three time points: at 3 weeks and at 6 months post randomization
  Generic QOL will be measured using Short-Form Health Survey-36 (SF-36) instrument. Physical and Mental Component Summary scores reflect physical and mental health status, respectively. To only take into account change in QOL related to DVT, at the 3 week visit, we will change the first sentence (i.e. stem) of the SF-36 questionnaire from 'over the past 4 weeks' to 'over the past 3 weeks'.
QOL (Quality of Life) score - VEINES-QOL | Three time points: at 3 weeks and at 6 months post randomization
  Venous disease-specific QOL will be assessed with VEINES-QOL, a 25-item self-completed measure. To only take into account change in QOL related to DVT, at the 3 week visit, we will change the first sentence (i.e. stem) of the VEINES-QOL questionnaire from 'over the past 4 weeks' to 'over the past 3 weeks'.
SAEs | baseline to 6 months post randomization
  Serious adverse events (SAE) will be defined as per the Health Canada definition. SAEs will be reported as required by local regulations, with copies sent to Health Canada, Therapeutic Product Directorate (Ottawa), Leo Pharma (maker of tinzaparin) and Bayer (maker of rivaroxaban). SAEs from baseline to 3 weeks and from 3 weeks to 6 months, including recurrent DVT, PE (Pulmonary Embolism), major bleeding and clinically relevant non-major bleeding, death will be assessed.
Rate of lost to follow-up | 6 months post randomization
  The number of patients randomized that do not attend (in person or over the phone) the 6-month follow-up visit; Patients who withdraw consent are not considered as lost to follow-up.

OTHER OUTCOMES:
Health Services Research Issues | 6 months post randomization
  QOL analyses will be conducted in the pilot study, as it is relevant to comprehensively evaluate chronic burdensome conditions like PTS. Utilities for health states will be derived from QOL measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Galanaud, MD, Principal Investigator — Sunnybrook Health Sciences Centre (Toronto, Ontario, Canada); Susan R Kahn, MD, Principal Investigator — Jewish General Hospital (Montreal, Quebec, Canada)
Locations (5):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montréal, Ontario
  - The Ottawa Hospital - Ottawa Hospital Research Institute (OHRI), Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makedonov I, Kahn SR, Galanaud JP. Prevention and Management of the Post-Thrombotic Syndrome. J Clin Med. 2020 Mar 27;9(4):923. doi: 10.3390/jcm9040923. PMID 32230912
- [Background] Kahn SR, Comerota AJ, Cushman M, Evans NS, Ginsberg JS, Goldenberg NA, Gupta DK, Prandoni P, Vedantham S, Walsh ME, Weitz JI; American Heart Association Council on Peripheral Vascular Disease, Council on Clinical Cardiology, and Council on Cardiovascular and Stroke Nursing. The postthrombotic syndrome: evidence-based prevention, diagnosis, and treatment strategies: a scientific statement from the American Heart Association. Circulation. 2014 Oct 28;130(18):1636-61. doi: 10.1161/CIR.0000000000000130. Epub 2014 Sep 22. No abstract available. PMID 25246013
- [Background] Hull RD, Townshend G. Long-term treatment of deep-vein thrombosis with low-molecular-weight heparin: an update of the evidence. Thromb Haemost. 2013 Jul;110(1):14-22. doi: 10.1160/TH12-12-0931. Epub 2013 Apr 25. PMID 23615656
- [Background] Kahn SR, Partsch H, Vedantham S, Prandoni P, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of post-thrombotic syndrome of the leg for use in clinical investigations: a recommendation for standardization. J Thromb Haemost. 2009 May;7(5):879-83. doi: 10.1111/j.1538-7836.2009.03294.x. Epub 2009 Jan 19. PMID 19175497
- [Derived] Makedonov I, Kahn S, Abdulrehman J, Schulman S, Delluc A, Gross PL, Galanaud JP. TILE pilot trial study protocol: Tinzaparin Lead-in to Prevent the Post-Thrombotic syndrome study protocol. BMJ Open. 2023 Oct 31;13(10):e064715. doi: 10.1136/bmjopen-2022-064715. PMID 37907305